CLINICAL TRIAL: NCT02687113
Title: Pre-procedure Planning for Radiofrequency Ablation Using the Automatic Fusion Images of the Registrated 3D CT or MR-US Scans: Preliminary Study
Brief Title: Pre-procedure Planning for Radiofrequency Ablation Using CT or MR/US Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-2361
Record Dates: First submitted 2016-02-11; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cancer
Keywords: ablation; fusion
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT/US fusion (Other): patients undergo routine conventional feasibility planning ultrasound, and clinical decision of RFA feasibility is made based on conventional planning ultrasound.
  Then additional planning ultrasound using CT/US fusion technique is immediately performed by the same operator, and clinical decision is made based on fusion imaging.
  Interventions: Device: CT/US fusion

INTERVENTIONS:
Device: CT/US fusion — Fusion of pre-RFA cross-sectional imaging (CT or MRI) and real-time USG using registration function of USG device.

SUMMARY:
The purpose of this study is to determine whether fusion technique of pre-radiofrequency ablation (RFA) cross-sectional imaging (CT or MR) and real-time ultrasonography would improve feasibility of RFA in patients with liver tumor in comparison with ultrasonography guidance alone.

DETAILED DESCRIPTION:
RFA is one of commonly used local therapies for primary or secondary liver tumors. For successful and safe procedure, safe route of electrode and lesion visibility are essential for RFA, and the conditions are usually evaluated on pre-RFA planning ultrasonography (USG). However, RFA is sometimes aborted due to limited sonic window of various cause and challenging identification of small isoechoic tumors or hepatocellular carcinomas among dysplastic nodules . Therefore, precise targeting and assuring safe route would be of clinical importance. In this preliminary study, investigators attempted to determine US and CT/MR fusion technique would be able to improve RFA feasibility in patients with liver tumors in comparison with conventional US alone technique.

ELIGIBILITY:
Inclusion Criteria: all conditions should be satisfied for inclusion.

* referred to Radiology in our institution for liver tumor RFA
* available pre-RFA liver CT or liver MR imaging within 6 weeks

Exclusion Criteria: patients with any of following condition should be excluded.

* any contraindication of liver RFA
* any patients who received treatment between pre-RFA imaging and planned RFA
* patients referred for palliative purpose.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
RFA feasibility rates on planning USG with/without fusion CT/MR and US | 10 minutes after finishing planning USG
  comparison of rates of RFA feasibility on conventional planning USG and on fusion planning USG

SECONDARY OUTCOMES:
Rate of tumor visibility on planning USG with/without fusion technique | 10 minutes after finishing planning USG
  comparison of tumor visibility (or detection) rates on planning USG on conventional planning USG and fusion planning USG
Number of patients with safety access route on planning USG with/without fusion technique | 10 minutes after finishing planning USG
  comparison of number of patients with presence/absence of safety access route, and the on two planning USGs

OTHER OUTCOMES:
Anticipated number of overlapping of RFA electrodes on planning USG with/without fusion technique | 30 minutes after finishing planning USG
  comparison of anticipated number of electrode overlapping on two planning USGs

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn SJ, Lee JM, Lee DH, Lee SM, Yoon JH, Kim YJ, Lee JH, Yu SJ, Han JK. Real-time US-CT/MR fusion imaging for percutaneous radiofrequency ablation of hepatocellular carcinoma. J Hepatol. 2017 Feb;66(2):347-354. doi: 10.1016/j.jhep.2016.09.003. Epub 2016 Sep 17. PMID 27650284